CLINICAL TRIAL: NCT05364775
Title: A Qualitative Study Exploring The Experiences Of International Nurses Working In The NHS
Brief Title: The Experiences of International Nurses
Status: Withdrawn | Type: Observational
Why Stopped: CI not pursuing study
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021NUR118
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Nurse's Role; Recruitment
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus Groups with International Nurses: It is anticipated that there will be four focus groups, each comprised of 6-8 participants
  Interventions: Other: Focus group
- Interviews with Nursing Staff: Interviews with qualified and unqualified staff who work with international nurses
  Interventions: Other: Focus group

INTERVENTIONS:
Other: Focus group — Focus group

SUMMARY:
The international mobility of the nursing workforce is increasing. One nurse out of every eight now works in a country where they were not born or trained. International nurses play a vital role in the NHS. This study focuses on the workplace experiences of international nurses who have trained outside of the EU. In recent years there have been increasing numbers of nurses from outside of the European Union (EU) registering to work in the UK, notwithstanding the number of nurses from European countries continues to decline as the UK prepares to leave the EU. There is currently a global shortage of nurses. Drivers for UK recruitment of international nurses are founded in shortages of nurses related to increased health care demand, emphasis on safe staffing levels, expenditure on agency nurses and too few commissions for nurse training places, meaning that not enough nurses are entering the NHS. These factors are further exacerbated by staff retention levels and high staff turnover. Nurses' motives to leave their home countries are complex, and gaps in our understandings remain. Possible drivers for migrating to the UK or "pull factors" may include career progression, postgraduate training opportunities, work environment, sensitive employment policies, and economic benefits which enable nurses to send money back to their home countries, while "push" factors have been identified as limited education, lack of health care resources, dangerous working conditions and political instability.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* International nurses recruited via the fellowship scheme and external recruitment agencies.
* International nurses who have trained in countries outside of the EU.
* International nurses who have been living in the UK between six months and two years.
* The international nurses will be employees of RWT

Phase 2

• Health Care Assistants and Qualified Nurses (Band 5-7) who alongside with international nurses.

Exclusion Criteria:

* International nurses who trained in the EU.
* International nurses who have lived in the UK for less than 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: International nurses, HCAs and Qualified Nurses who fit the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
The findings of the study will identify factors influencing the experiences of internationally recruited nurses working in the NHS | 6 months
  To identify factors influencing the experiences of internationally recruited nurses working in the NHS
The findings may also suggest ways in which RWT can further support international nurses to ensure successful professional and social integration. | 6 months
  To suggest ways in which RWT can further support international nurses to ensure successful professional and social integration.
This support could be put in place to benefit the local teams, patients and services. | 6 months
  To benefit local teams, patients and services.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom